CLINICAL TRIAL: NCT00194584
Title: Building on Family Strengths: An Educational Program for Parents of Children With On-Going Health Care Needs
Brief Title: Childhood Chronic Illness: An Educational Program for Parents of Children With On-Going Health Care Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Gail Kieckhefer, PhD, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 04-0564-01; 1R01HS013384-04 (AHRQ)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Illness
Keywords: children; chronic illness; parent education; parent support
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: 7 week Building on Family Strengths Program
- 0 (No Intervention)

INTERVENTIONS:
Behavioral: 7 week Building on Family Strengths Program — Parents in intervention group attend a 2 hr class for seven weeks. These classes provide information, time for discussion and creation of an action plan for the parent to complete in the intervening week.
  Arms: 1

SUMMARY:
The long-term goal of this research is to strengthen parents' abilities to manage the complexities of childhood chronic illness. To achieve this goal, the team of parents, health care professionals, and researchers proposes the following specific aim:

* Develop, implement, and test a unique psycho-educational program, Living with Childhood Chronic Illness (the Program), for effectiveness with parents of children who have chronic illnesses.

The investigators propose the following hypotheses:

At both 6 and 12 month follow-up points, parents taking part in the intervention, in contrast to control parents, will have:

1. Greater perceived self-efficacy regarding their ability to manage the child's chronic condition;
2. Greater parental ability to involve their child in shared management activities;
3. Greater parental ability to cope at 6 and 12 months following the end of the intervention;
4. Greater emotional health; and
5. Greater parental perceived family quality of life.

DETAILED DESCRIPTION:
Parents will enroll in the study by contacting the study number: 206-987-1000 or by sending an email message to family.strengths@seattlechildrens.org. They will complete a survey taking no more than 60 minutes. Parents will then be randomized to either take the class immediately or be in the control group which can take the class in 12 months. At the end of 6 and 12 months all the participants again take the survey.

Classes are 7 weeks in length, 2 hours each and are offered at various locations throughout the Greater Seattle area.

ELIGIBILITY:
Inclusion Criteria:

* Child 2-11 years of age, with diagnosed chronic illness
* Parent at least 18 years of age, able to speak and read English at 4th grade level and able to attend a 7 week two-hour class program

Exclusion Criteria:

* Child in active hospice treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2004-10; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
depressive symptoms | 6, and 12 months

SECONDARY OUTCOMES:
self-efficacy | 6 and 12 months
parent-child shared management | 6, and 12 months
coping | 6, and 12 months
quality of life | 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gail M Kieckhefer, PhD, Principal Investigator — University of Washington